CLINICAL TRIAL: NCT01011660
Title: Phase 4 Study of Effects of ARB Compared With Diuretics in Hypertension Patients With High Cardiovascular Risks
Brief Title: Effects of Angiotensin II Receptor Blocker Compared With Diuretics in High-risk Hypertensive Patients
Acronym: CHIEF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Ma Liyuan, Dr, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 115
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Essential Hypertension
Keywords: hypertension; cardiovascular risk factors; drugs intervention; lipid-lowering therapy; 50-79 years of age; sign; the informed; consent; forms
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Amlodipine; Telmisartan; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A,1,IV (Active Comparator): A means active; 1 means Amlodipine+Amiloride Compound; IV means phase IV
  Interventions: Drug: Amlodipine, Telmisartan, Amiloride Compound , Simvastatin
- A,2,IV (Active Comparator): A means active; 2 means Amlodipine+Telmisartan; IV means phase IV
  Interventions: Drug: Amlodipine, Telmisartan, Amiloride Compound , Simvastatin
- A,3,IV (Active Comparator): A means active; 3 means Amlodipine+Amiloride Compound with or no Simvastatin; IV means phase IV
  Interventions: Drug: Amlodipine, Telmisartan, Amiloride Compound , Simvastatin
- A,4,IV (Active Comparator): A means active; 4 means Amlodipine+Telmisartan with or no Simvastatin; IV means phase IV
  Interventions: Drug: Amlodipine, Telmisartan, Amiloride Compound , Simvastatin

INTERVENTIONS:
Drug: Amlodipine, Telmisartan, Amiloride Compound , Simvastatin — Amlodipine; Telmisartan; Amiloride Compound; Simvastatin
  Other Names: CHIEF

SUMMARY:
The aim of the study is to investigate the optimized treatment strategy of hypertension, so as to make more patients to reach the blood pressure goals and to reduce cardio-cerebrovascular events. Objective and Methods: Patients are eligible for inclusion in the study if they are essential hypertension, 50-79 years of age with at least one cardiovascular risk factor and sign the informed consent forms. This project is a multi-centre, prospective randomized,，openlabel blind-endpoint evaluation controlled (PROBE) trial. 12000 patients will be randomly assigned to either of low-dose Amlodipine+Telmisartan group or Amlodipine+ diuretics group. Among those patients with serum cholesterol between 4.0-6.1mmol/L, they will be also randomized into small dose of statin-based regimen or standard management regimen; Patients will also randomly assigned to intensive lifestyle intervention group or standard intervention group according to the community area where the patients in.

DETAILED DESCRIPTION:
This study is aimed to observe the main outcome (stroke, myocardial infarction and death from cardiovascular disease) differences between different groups.

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension
* 50-79 years old
* with at least one of the cardiovascular risk factor
* sign consent forms

Exclusion Criteria:

* secondary hypertension
* attack of cerebrovascular events or myocardial infarction within recent 3 months
* coexistence of severe cardiomyopathy, rheumatic or congenital heart diseases
* unstable angina
* severe hepatopathy or nephropathy (ALT elevation > 2 fold or serum creatinine > 2.5mg/dl)
* malignant tumor
* gout
* women taking contraceptives or with pregnancy
* allergic history to the research drugs
* validated contradiction to the research drugs
* participating in other clinical trials
* unable for long-term follow-up or poor compliance
* unsuitable for clinical trial at the discretion of doctors in charge

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13542 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary study outcomes are composite of non-fatal stroke, non-fatal myocardial infarction and cardiovascular death. | 3-4 years

SECONDARY OUTCOMES:
All cardiovascular events；all-cause death, hospitalization for angina pectoris, coronary revascularization, aortic dissection, cerebrovascular disease, heart failure, renal insufficiency, tumor, new onset of atrial fibrillation and diabetes mellitus | 3-4 years

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wang, Professor, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Wang Wen, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ma L, Wang W, Zhao Y, Zhang Y, Deng Q, Liu M, Sun H, Wang J, Liu L. Combination of amlodipine plus angiotensin receptor blocker or diuretics in high-risk hypertensive patients: a 96-week efficacy and safety study. Am J Cardiovasc Drugs. 2012 Apr 1;12(2):137-42. doi: 10.2165/11598110-000000000-00000. PMID 22329591